CLINICAL TRIAL: NCT04423783
Title: Testing a Gamified App to Reduce Avoidance and Fear of Spiders in Spider Phobia
Brief Title: Gamification in the Treatment of Spider Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anke Haberkamp (Other)
Responsible Party: Sponsor-Investigator, Anke Haberkamp, Principal Investigator, Philipps University Marburg
Organization: Philipps University Marburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GaSpPh
Record Dates: First submitted 2020-05-14; First posted 2020-06-09 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Spider Phobia
Keywords: Gamification; Anxiety Disorder; Avoidance; App
MeSH Terms: conditions — Arachnophobia; Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spider gamification app (Experimental): Participants play the spider gamification app twice a day for 7 days
  Interventions: Behavioral: 7-day exposure therapy via self-developed app according to (Haberkamp et al., submitted)
- Online exposure + spider gamification app (Experimental): Participants receive a therapist-guided one-session online exposure therapy and play the spider gamification app twice a day for 7 days
  Interventions: Behavioral: 7-day exposure therapy via self-developed app according to (Haberkamp et al., submitted); Behavioral: Therapist-guided one-session online exposure therapy according to (Öst, 1989)
- Online exposure + non-spider gamification app (Active Comparator): Participants receive a therapist-guided one-session online exposure therapy and play a non-spider gamification app twice a day for 7 days
  Interventions: Behavioral: Therapist-guided one-session online exposure therapy according to (Öst, 1989)

INTERVENTIONS:
Behavioral: 7-day exposure therapy via self-developed app according to (Haberkamp et al., submitted) — Confrontation with spiders via gamified app
  Other Names: Spider Gamification App
  Arms: Online exposure + spider gamification app; Spider gamification app
Behavioral: Therapist-guided one-session online exposure therapy according to (Öst, 1989) — Massed exposure therapy over the course of one single session, applied in a remote-online context
  Other Names: Online exposure
  Arms: Online exposure + non-spider gamification app; Online exposure + spider gamification app

SUMMARY:
Mobile applications are more and more considered when implementing programs for treating mental disorders. The study aims to reduce avoidance and fear of spiders in spider-fearful individuals by combining exposure principles with gamification elements (e.g. narrative background, level progression, points, feedback). We investigate the efficacy of the gamified app in a remote online-therapy context.

ELIGIBILITY:
Inclusion Criteria:

Participants must

* be 18 years or older,
* SPQ score ≥ 14
* BDI-II score ≤ 18

Exclusion Criteria:

Participants will be deemed ineligible if they do not meet the above inclusion criteria or

* are allergic to spiders or bee stings,
* are currently undergoing psychotherapeutic and/or psychopharmacological treatments,
* are experiencing current psychosis, mania, or substance abuse, or
* successfully complete 8 or more of 12 possible BAT steps at baseline (to ensure that participants are indeed spider fearful)
* are at higher risk from Covid-19 or
* participated in a pilot study in 2019.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in avoidance behavior (Behavioral Approach Task; BAT) | Baseline; (after one-session exposure if applied); Post-treatment (1-week after baseline); 3-week follow-up (4-weeks after baseline)
  Scores range from 0 ("participant refuses to enter the room with spider") to 12 ("participant holds the spider at least for 20 sec").
Change in spider fear (Spider Phobia Questionnaire; SPQ) | Baseline; Post-treatment (1-week after baseline); 3-week follow-up (4-weeks after baseline)
  The scale ranges from 0-31. High scores reflect high subjective levels and low scores low subjective levels of spider fear.
Change in spider fear: Spider-Anxiety Questionnaire (FAS) | Baseline; Post-treatment (1-week after baseline); 3-week follow-up (4-weeks after baseline)
  The scale ranges from 0-108. High scores reflect high subjective levels and low scores low subjective levels of spider fear.

SECONDARY OUTCOMES:
Change in disgust before and after playing the app | Before starting and immediately after completing the game
  Seven-point rating scale scoring from 0 to 6: high scores reflect high levels and low scores low levels of experienced disgust; participants play twice a day (between 8 - 11 am and 4 - 7 pm); ratings are part of the app
Change in arousal before and after playing the app | Before starting and immediately after completing the game
  Seven-point rating scale scoring from 0 to 6: high scores reflect high levels and low scores low levels of experienced arousal; participants play twice a day (between 8 - 11 am and 4 - 7 pm); ratings are part of the app
Change in anxiety before and after playing the app | Before starting and immediately after completing the game
  Seven-point rating scale scoring from 0 to 6: high scores reflect high levels and low scores low levels of experienced anxiety; participants play twice a day (between 8 - 11 am and 4 - 7 pm); ratings are part of the app

OTHER OUTCOMES:
Beck Depression Inventory II (BDI-II) | Baseline, Post-treatment (1-week after baseline); 3-week follow-up (4-weeks after baseline)
  Measures severity of depression; The scale ranges from 0-63: 0-13 minimal depressive symptoms; 14-19 mild symptoms; 20-28 moderate symptoms; 29-63 severe symptoms.
Brief Symptom Inventory (BSI) | Baseline, Post-treatment (1-week after baseline); 3-week follow-up (4-weeks after baseline)
  Measures clinically relevant psychological symptoms.
German version of the Client Satisfaction Questionnaire (CSQ-8) | (after one-session exposure if applied), Post-treatment (1-week after baseline); 3-week follow-up (4-weeks after baseline)
  Standardised satisfaction measurement
Mobile Application Rating Scale (MARS) | Post-treatment (1-week after baseline)
  Questionnaire assessing the quality of new user-oriented health applications

CONTACTS AND LOCATIONS:
Overall Officials: Anke Haberkamp, PhD, Principal Investigator — Philipps University Marburg
Locations (2):
- Germany (2):
  - Philipps University Marburg, Marburg
  - Philipps-University Marburg Clinical Psychology and Psychotherapy, Marburg

IPD SHARING:
Plan to Share IPD: Yes
Share anonymized IPD via a general-purpose open-access repository
Time Frame: end of the study; unlimited
Access Criteria: open-access